CLINICAL TRIAL: NCT02565667
Title: A Prospective Randomized Clinical Study for Transanal Double Purse-string Rectal Anastomosis Preformed With KOL Stapler
Brief Title: A Prospective Clinical Study for Transanal Double Purse-string Rectal Anastomosis Preformed With KOL Stapler
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, LI XIN-XIANG, professor of colorectal surgery, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FudanKOL
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Rectal Neoplasms
Keywords: low rectal carcinoma; anastomosis; anterior rectal resection
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KOL group (Experimental): KOL stapler was used for rectal anastomosis
  Interventions: Device: KOL
- traditional stapler group (Active Comparator): traditional stapler was used for rectal anastomosis
  Interventions: Device: traditional staple

INTERVENTIONS:
Device: KOL — KOL staple was used for rectal anastomosis
  Arms: KOL group
Device: traditional staple — traditional staple was used for rectal anastomosis
  Arms: traditional stapler group

SUMMARY:
The most challenge for the surgery of low rectal carcinoma was whether to perform low anterior resection (LAR) and preserve anal function improving the quality of life for patients, for which anastomotic leak is a great obstacle with about 5-10% incidence in reported literature. Up to now, kinds of surgical devices have been employed to reduce anastomotic leak rate after LAR. Most of these anastomotic devices could not resolve the problem of "dog ear" phenomena. In the present clinical trial, the investigators use a double purse-string rectal anastomosis with KOL staple in laparoscopic anterior rectal resection for low or ultra-low rectal carcinoma, which will resolve the problem of dog ear. The investigators aim to demonstrate the safety, effectiveness of this procedure and establish a standard method for laparoscopic (ultra-)low anterior rectal resection.

DETAILED DESCRIPTION:
About 5-10% of patients receiving low rectal resection using traditional anastomosis occurred anastomotic leak, risk factors for which included patient related (age, gender, tumor distance from the anal verge), hypoproteinemia, diabetes mellitus, etc), procedure related (emergency) and technical related (one stapler, double stapler or handsewn).

Anastomotic leak caused prolonged hospital stay, delayed post-operative adjuvant radiochemotherapy and need of stoma in some cases. Besides, anastomotic leak was reported to be associated with increased local recurrence rate. Thus, it's of great importance to develop new surgical devices to prevent "dog ear" problem and reduce the anastomotic leak rate.

Double stapled pursestring anastomosis was the one of the most widely used methods in lower rectal resection. One major problem of this procedure was creating one or double side "dog ear" phenomenon (Dis Colon Rectum. 2000 Apr;43(4):522-5. Fig 1). This weak spot was theoretically responsible for post-operative anastomotic leak as demonstrated by animal experiments and clinical practice.

In this clinical trial, we used a transanal double purse-string rectal anastomosis preformed with KOL stapler for lower rectal resection. This procedure would resolve the dog ear problem through circular anastomosis taking care that the anastomotic site contained only gut tissues without any staples. We aim to demonstrate the safety, effectiveness of this procedure and establish a standard method for laparoscopic (ultra-)low anterior rectal resection.

ELIGIBILITY:
Inclusion Criteria:

1. pathological confirmed rectal adenocarcinoma
2. less than 10 cm of distal tumor margin from the anal edge
3. less than 4 cm of maximum tumor diameter and less than 1/2 of circumference diameter
4. tumor stage earlier than cT1-3N0M0 before surgery or that following neoadjuvant radiochemotherapy
5. normal defecation function (Wexner score < 4)
6. open or laparoscopic operation

Exclusion Criteria:

1. recurrent cases
2. emergency including obstruction, bleeding or perforation
3. severe abdominal adhesions
4. severe malnutrition can not be improved before surgery
5. can not tolerate to surgery due to severe comorbidities of heart, lung, liver or kidney
6. refractory hypoproteinemia or diabetes mellitus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
anastomotic leak rate | 30 days since the date of surgery
  percentage of patients occuring anastomotic leak within 30 days since surgery

SECONDARY OUTCOMES:
post-operative anal function | within one year since the date of surgery
30-day mortality rate | within 30 days since the date of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Li Xin-Xiang, M.D & Ph.D., Study Director — Shanghai Cancer Center, Fudan University, #270 Dong An Road, Shanghai, 200030
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Midura EF, Hanseman D, Davis BR, Atkinson SJ, Abbott DE, Shah SA, Paquette IM. Risk factors and consequences of anastomotic leak after colectomy: a national analysis. Dis Colon Rectum. 2015 Mar;58(3):333-8. doi: 10.1097/DCR.0000000000000249. PMID 25664712
- [Background] Espin E, Ciga MA, Pera M, Ortiz H; Spanish Rectal Cancer Project. Oncological outcome following anastomotic leak in rectal surgery. Br J Surg. 2015 Mar;102(4):416-22. doi: 10.1002/bjs.9748. Epub 2015 Jan 26. PMID 25619499
- [Background] Trencheva K, Morrissey KP, Wells M, Mancuso CA, Lee SW, Sonoda T, Michelassi F, Charlson ME, Milsom JW. Identifying important predictors for anastomotic leak after colon and rectal resection: prospective study on 616 patients. Ann Surg. 2013 Jan;257(1):108-13. doi: 10.1097/SLA.0b013e318262a6cd. PMID 22968068
- [Background] Morse BC, Simpson JP, Jones YR, Johnson BL, Knott BM, Kotrady JA. Determination of independent predictive factors for anastomotic leak: analysis of 682 intestinal anastomoses. Am J Surg. 2013 Dec;206(6):950-5; discussion 955-6. doi: 10.1016/j.amjsurg.2013.07.017. Epub 2013 Sep 24. PMID 24070663
- [Background] Mirnezami A, Mirnezami R, Chandrakumaran K, Sasapu K, Sagar P, Finan P. Increased local recurrence and reduced survival from colorectal cancer following anastomotic leak: systematic review and meta-analysis. Ann Surg. 2011 May;253(5):890-9. doi: 10.1097/SLA.0b013e3182128929. PMID 21394013
- [Background] Roumen RM, Rahusen FT, Wijnen MH, Croiset van Uchelen FA. "Dog ear" formation after double-stapled low anterior resection as a risk factor for anastomotic disruption. Dis Colon Rectum. 2000 Apr;43(4):522-5. doi: 10.1007/BF02237198. PMID 10789750